CLINICAL TRIAL: NCT07380334
Title: An Open Label, Multicenter Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-1049 Injection in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-1049 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1049-101
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SHR-1049 Group - Queue 1 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection
- SHR-1049 Group - Queue 2 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection
- SHR-1049 Group - Queue 3 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection
- SHR-1049 Group - Queue 4 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection
- SHR-1049 Group - Queue 5 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection
- SHR-1049 Group - Queue 6 (Experimental): Specified dose on specified days.
  Interventions: Drug: SHR-1049 Injection

INTERVENTIONS:
Drug: SHR-1049 Injection — SHR-1049 injection.

SUMMARY:
This study is a multicenter, open label, dose exploration/efficacy extension Phase I clinical trial aimed at evaluating the safety, tolerability, pharmacokinetics and efficacy of SHR-1049 injection in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study, sign the informed consent form, have good compliance, and can cooperate with follow-up;
2. Age range of 18-75 years old (including 18 and 75 years old, calculated on the day of signing informed consent), both male and female are eligible;
3. Dose exploration stage: Participants with advanced or metastatic solid tumors diagnosed by tissue or cytological pathology who have failed standard treatment (disease progression or toxicity intolerance) or have no effective standard treatment;
4. Stage of efficacy extension: Late stage or metastatic solid tumors diagnosed by tissue or cytological pathology;
5. Able to provide sufficient fresh or archived tumor tissue specimens for third-party central laboratories designated by the sponsor to test expression levels; For participants who are unable to provide tumor tissue samples, the decision to enroll will be made after joint evaluation by the researchers and the sponsor;
6. At least one measurable lesion that meets RECIST v1.1 criteria; Lesions that have undergone local treatment, if there is clear evidence of significant progression after treatment, can be selected as target lesions;
7. ECOG PS score: 0 to 1;
8. Expected survival period ≥ 12 weeks;
9. The function of important organs meets the requirements;
10. Female participants with fertility must have a negative serum HCG test within 7 days prior to their first medication and must be non lactating; Female participants with fertility must agree to use contraception and avoid egg donation for a period of 7 months from the signing of the informed consent form until the last administration of the investigational drug; Male participants whose partners are fertile women must agree to contraception and avoid donating sperm for a period of 4 months from the signing of the informed consent form until the last administration of the investigational drug.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis; Participants with a history of meningeal metastasis or current meningeal metastasis;
2. Imaging shows tumor invasion of large blood vessels or unclear boundary with blood vessels; Or it may be determined by researchers that the participant's tumor has a high possibility of invading important blood vessels and causing fatal massive bleeding during treatment;
3. Previous or concurrent presence of other malignant tumors;
4. Chest effusion, pericardial effusion, or abdominal effusion that is accompanied by clinical symptoms, difficult to control, or moderate or above; If fluid drainage is performed (excluding diagnostic puncture surgery), those who have been stable for at least 2 weeks after drainage can be included in the group;
5. Interstitial pneumonia/interstitial lung disease, non infectious pneumonia (such as radiation pneumonitis) that previously required steroid treatment; Currently present or suspected of having interstitial pneumonia/interstitial lung disease, non infectious pneumonia, or other active pneumonia; Severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, and other lung damage occurred within 6 months prior to the first use of medication; Individuals with active pulmonary tuberculosis;
6. Accompanied by poorly controlled or severe cardiovascular disease;
7. Within one month prior to the first medication, there has been a bleeding event with NCI-CTCAE v5.0 grade ≥ 2;
8. Those who have experienced or are expected to experience gastrointestinal perforation or fistula, tracheal fistula, urethral fistula, or abdominal abscess within 3 months before the first medication;
9. Symptoms and signs of gastrointestinal obstruction or gastrointestinal obstruction within 3 months prior to the first use of medication;
10. Participants who have experienced a severe infection within one month prior to their first medication;
11. History of immunodeficiency, including HIV test positive, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; Participants known to have active hepatitis or active hepatitis C;
12. Patients who have previously undergone surgery (excluding diagnostic surgery), radiotherapy, local treatment, chemotherapy, macromolecular targeted therapy, anti-tumor immunotherapy, and have completed treatment (last medication) less than 4 weeks after the first medication; Small molecule targeted drugs (including other oral targeted drugs used in clinical trials) with less than 5 half lives or 4 weeks (whichever is shorter) between the last dose and the first dose;
13. Previously received drug treatment with the same mechanism as the experimental drug;
14. According to NCI-CTCAE v5.0 classification, those whose toxicity caused by previous anti-tumor therapy has not yet recovered to ≤ grade 1;
15. Individuals known to be allergic to any component or other antibody drugs of SHR-1049 product;
16. Those who have received attenuated live vaccine within 4 weeks before the first administration or are likely to receive attenuated live vaccine during treatment and within 60 days after the last administration;
17. According to the researcher's judgment, there are other factors that may affect the research results or force the termination of this study midway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of dose-limiting toxicity (DLT). | Expected results within one year.
  The first dosing cycle after each subject's enrollment is the DLT observation period.
Adverse events (AEs). | Approximately 12 months after the last patient enrolled.
  Continuous observation from each participant's knowledge until the end of the safety follow-up period.
Serious adverse events (SAEs). | Approximately 12 months after the last patient enrolled.
  Continuous observation from each participant's knowledge until the end of the safety follow-up period.
Maximum tolerated dose (MTD). | Plan to obtain results within 10 months of the first dose ramp up.
  Based on the preliminary data summary evaluation, it is estimated that after completing the dose group ramping up and expanding the efficacy of 1-2 cohorts into the group with preliminary efficacy results, corresponding results can be obtained.
Recommended dose for phase II clinical study (RP2D). | Plan to obtain results within 20 months of the first dose ramp up.
  Based on the preliminary data summary evaluation, it is estimated that after completing the dose group ramping up and expanding the efficacy of 1-2 cohorts into the group with preliminary efficacy results, corresponding results can be obtained.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator - Blood drug concentration. | The plan is to complete all evaluations within 2 years.
  The plan is to conduct an evaluation within 4 weeks after each dose escalation and within 4 weeks after each dose expansion. The PK evaluation of efficacy expansion needs to be evaluated based on specific preliminary data as appropriate.
Immunogenic indicator - Anti-drug antibody (ADA) levels. | The plan is to complete all evaluations within 2 years.
  The plan is to conduct an evaluation within 4 weeks after each dose escalation and within 4 weeks after each dose expansion. The ADA evaluation of efficacy expansion needs to be evaluated based on specific preliminary data as appropriate.
Effectiveness indicator - Researchers evaluated objective response rate (ORR). | Approximately 12 months after the last patient enrolled.
  After the first medication, imaging examinations should be conducted every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (±7 days) thereafter, and follow-up should be continued until the subject's imaging progress.
Effectiveness indicator - Researchers evaluated duration of response (DoR). | Approximately 12 months after the last patient enrolled.
  After the first medication, imaging examinations should be conducted every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (±7 days) thereafter, and follow-up should be continued until the subject's imaging progress.
Effectiveness indicator - Researchers evaluated disease control rate (DCR). | Approximately 12 months after the last patient enrolled.
  After the first medication, imaging examinations should be conducted every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (±7 days) thereafter, and follow-up should be continued until the subject's imaging progress.
Effectiveness indicator - Researchers evaluated progression free survival (PFS). | Approximately 12 months after the last patient enrolled.
  After the first medication, imaging examinations should be conducted every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (±7 days) thereafter, and follow-up should be continued until the subject's imaging progress.
Effectiveness indicator - Researchers evaluated overall survival (OS) based on the RECIST v1.1 evaluation criteria for solid tumor treatment efficacy. | Approximately 12 months after the last patient enrolled.
  After the first medication, imaging examinations should be conducted every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (±7 days) thereafter, and follow-up should be continued until the subject's imaging progress.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided